CLINICAL TRIAL: NCT05436509
Title: CD19/79b Bi-specific CAR-T Cells Targeting B Cell Malignancies
Brief Title: CD19/79b Bi-specific CAR-T Cell Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-22009
Record Dates: First submitted 2022-06-22; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: B Cell Malignancies
Keywords: CAR-T; B cell Malignancies; CD19; CD79b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bi-4SCAR-CD19/79b T Cell Therapy for CD19 and/or CD79b positive B cell malignancies (Experimental)
  Interventions: Biological: bi-4SCAR CD19/79b T cells

INTERVENTIONS:
Biological: bi-4SCAR CD19/79b T cells — Infusion of bi-4SCAR-CD19/79b T cells at 10^6 cells/kg body weight via IV

SUMMARY:
The purpose of this study is to assess the feasibility, safety and efficacy of CD19/79b bi-specific CAR-T cell therapy in patients with CD19 and/or CD79b positive B cell malignancies. Another goal of the study is to learn more about the safety and function of the anti-CD19/79b bi-specific CAR-T cells and their persistency in patients.

DETAILED DESCRIPTION:
Patients with refractory and/or recurrent B cell malignancies have poor prognosis despite complex multimodal therapy. Despite impressive progress, more than 50% of patients treated with CD19-targeting chimeric antigen receptor T cells (CAR19) experience progressive disease. Further, more than 40% patients with progressive large B cell lymphoma (LBCL) experienced reduced or lost expression of CD19 on the tumor cells after CAR19 treatment; low surface CD19 density before treatment was associated with progressive disease. Therefore, novel curative approaches are needed. The investigation attempts to use genetically modified T cells to express a 4th generation lentiviral anti-CD19/79b bi-specific CAR (bi-4SCAR-CD19/79b). The CAR molecules enable the T cells to recognize and kill tumor cells through the recognition of a surface antigen, CD19 or CD79b, which is expressed at high levels on tumor cells but not at significant levels on normal tissues.

CD79b is a B cell surface antigen, which is a component of B cell receptor. CD79b is up-regulated in more than 90% of B-cell lymphomas. Recent studies have shown that CD79b CAR-T cells have potential in targeting B-cell lymphomas. In addition, several immunotherapy drugs based on targeting CD79b have been reported worldwide. The CD79b specific CAR-T cells with binding moiety of CD79b specific scFv exhibited a high affinity and antitumor effect against CD79b+ tumor cells.

A potential strategy to prevent relapse due to antigen escape is to infuse T-cells capable of recognizing multiple antigens. To overcome tumor escape of single target antigen and enhance in vivo CAR-T efficacy, a novel bi-specific CD19/79b CAR-T therapy regimen is developed to include booster and consolidation CAR-T applications to target highly-refractory B cell cancer. The aim is to evaluate safety and long term efficacy of the bi-CAR-T therapy strategy in CD19 and/or CD79b positive cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. age older than 6 months.
2. malignant B cell surface expression of CD19 or CD79b molecules.
3. the KPS score over 80 points, and survival time is more than 1 month.
4. greater than Hgb 80 g/L.
5. no contraindications to blood cell collection.

Exclusion Criteria:

1. accompanied with other active diseases and difficult to assess patient response.
2. bacterial, fungal, or viral infection, unable to control.
3. living with HIV.
4. active HBV or HCV infection.
5. pregnant and nursing mothers.
6. under systemic steroid treatment within a week of the treatment.
7. prior failed CD19 and CD79b CAR-T treatment.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of fourth generation bi-4SCAR-CD19/79b T cells in patients with B cell malignancies | 12 weeks
  Safety of fourth generation bi-4SCAR-CD19/79b T cells in patients with B cell malignancies using CTCAE 4 standard to evaluate the level of adverse events standard to evaluate the level of adverse events

SECONDARY OUTCOMES:
Anti tumor activity of fourth generation bi-4SCAR-CD19/79b T cells in patients with relapsed or refractory B cell malignancies | 1 year
  Scale of CAR copies (for efficacy)
Anti tumor activity of fourth generation bi-4SCAR-CD19/79b T cells in patients with relapsed or refractory B cell malignancies | 1 year
  Scale of leukemic cell burden (for efficacy)

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No